CLINICAL TRIAL: NCT02813408
Title: Prospective Multi-country Observational Study to Investigate the Impact of Abiraterone Acetate and Enzalutamide on Health-related Quality of Life, Patient-reported Outcomes, and Medical Resource Use in Metastatic Castration-resistant Prostate Cancer Patients
Brief Title: A Study to Investigate the Impact of Abiraterone Acetate and Enzalutamide on Health-related Quality of Life, Participant-Reported Outcomes, and Medical Resource Use in Metastatic Castration-resistant Prostate Cancer Participants
Acronym: AQUARiUS
Status: Completed | Type: Observational
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108141; 212082PCR4039 (Other: Janssen Pharmaceutica N.V., Belgium)
Record Dates: First submitted 2016-05-24; First posted 2016-06-27 (Estimated); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with Prostate Cancer (abiraterone acetate): Participants with metastatic castration resistant prostate cancer (mCRPC) will receive abiraterone acetate at the discretion of his treating physician.
- Participants with Prostate Cancer (enzalutamide): Participants with metastatic castration resistant prostate cancer (mCRPC) will receive enzalutamide at the discretion of his treating physician.

SUMMARY:
The purpose of this observational study of metastatic castration-resistant prostate cancer (mCRPC) participants is to explore whether or not there are differences between participants treated with abiraterone acetate and enzalutamide on the health-related quality of life (HRQoL), Fatigue, Pain, Cognitive function and medical resource use (MRU).

ELIGIBILITY:
Inclusion Criteria:

* Male 18 years of age or older
* Participant with histologically or cytologically confirmed diagnosis of adenocarcinoma of the prostate
* Participant with documented metastatic prostate cancer
* Participant with documented castration resistance with progression of prostate cancer on androgen deprivation therapy (ADT)
* Participant who will be initiated on either abiraterone acetate or enzalutamide for the treatment of metastatic castration-resistant prostate cancer (mCRPC) that is asymptomatic or mildly symptomatic (per physician's evaluation) after failure of ADT at the time of treatment initiation
* Participants who signed a participation agreement or Informed consent form (ICF) per local regulations
* The treatment decision (abiraterone acetate or enzalutamide) by the treating physician must have been taken before enrollment into the study
* Baseline patient-reported outcomes (PROs) must be captured before the first administration of abiraterone acetate or enzalutamide.

Exclusion Criteria:

* Patient who has received any chemotherapy/cytotoxic agent to treat their mCRPC before abiraterone acetate or enzalutamide initiation; or ; treat their metastatic hormone-sensitive prostate cancer (mHSPC) <12 months prior to abiraterone acetate or enzalutamide initiation.
* Participant who is not capable of completing a patient survey
* Participant who has received or is currently receiving abiraterone acetate or enzalutamide
* Patient receiving an investigational treatment for prostate cancer of any kind before or at the time of initiation of abiraterone acetate or enzalutamide
* Participant who is currently included in other observational studies with abiraterone acetate sponsored by Janssen

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who will initiate treatment with abiraterone acetate or enzalutamide at study entry will be observed.
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2016-05-03 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2018-03-21 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of Life (HRQoL) | 12 months
Fatigue (BFI-SF) | 12 months
  Brief Fatigue Inventory-Short Form (BFI-SF) assess the severity of fatigue and the impact of fatigue on daily functioning. BFI-SF is a 4 item questionnaire. Each item is assessed on a 11point scale, ranges from 0 (No Fatigue) to 10 (As bad as you can imagine). Average from all 4 items will be used to derive the final score.
Pain (BPI-SF) | 12 months
  Brief Pain Inventory-Short Form (BPI-SF) measures severity of pain, impact of pain on daily function, locations of pain, pain medications, and amount of pain relief in the past 24 hours or the past week. The BPI-SF includes 4 items measuring the intensity of pain which make up the pain intensity sub scales, assessed using 11 point numerical rating scales from "0"= no pain to "10" = pain as bad as you can imagine; 7 items that assess how much pain has interfered with 7 daily activities which make up the pain interference sub scale, assessed on a scale of 0, "Does not interfere" to 10, "completely interferes." This sub scale is typically scored as the mean of the 7 interference items; An additional item on the extent of pain relief.
Cognitive Function (FACT-Cog) | 12 months
  The Functional Assessment of Cancer Therapy-Cognitive (FACT-Cog) is a validated, 37 item, subjective neuro-psychological instrument designed to evaluate cancer participants perceived cognitive deterioration on their quality of life. The FACT-Cog is composed of 37 single items ranging from 04. Based on these single items 4 sub scales are calculated as perceived Cognitive Impairments (20 items; score range 0-80), impact On QOL (4 items; score range 0-16), comments From Others (4 items; score range 0-16), perceived Cognitive Abilities (9 items; score range 0-36).
Medical Resource Use (MRU) | 6 months prior to baseline until the end of the follow-up period (up to 18 months)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V., Belgium Clinical Trial, Study Director — Janssen Pharmaceutica N.V., Belgium
Locations (26):
- Denmark (3):
  - Holstebro
  - Næstved
  - Odense
- France (13):
  - Besançon
  - Beuvry
  - Bordeaux
  - Challes-les-Eaux
  - Chalon-sur-Saône
  - Dijon
  - Lyon
  - Marseille
  - Paris
  - Quimper
  - Saint-Mandé
  - Strasbourg
  - Toulouse
- United Kingdom (10):
  - Berkshire
  - Birmingham
  - Bolton
  - Derby
  - Glasgow
  - Lancaster
  - Middlesbrough
  - Oldham
  - Sutton
  - Wolverhampton

REFERENCES:
- [Derived] Thiery-Vuillemin A, Poulsen MH, Lagneau E, Ploussard G, Birtle A, Dourthe LM, Beal-Ardisson D, Pintus E, Trepiakas R, Lefresne F, Lukac M, Van Sanden S, Pissart G, Reid A; AQUARiUS Investigators. Impact of Abiraterone Acetate plus Prednisone or Enzalutamide on Patient-reported Outcomes in Patients with Metastatic Castration-resistant Prostate Cancer: Final 12-mo Analysis from the Observational AQUARiUS Study. Eur Urol. 2020 Mar;77(3):380-387. doi: 10.1016/j.eururo.2019.09.019. Epub 2019 Oct 5. PMID 31594705